CLINICAL TRIAL: NCT04289012
Title: HELicobacter Pylori Screening to Prevent Gastrointestinal Bleeding in Patients With Acute Myocardial Infarction Pilot Study
Brief Title: HELicobacter Pylori Screening in Patients With Acute Myocardial Infarction Pilot Study
Acronym: HELPpilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Robin Hofmann, MD, PhD. Principal investigator., Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HELP-MI pilot
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI
Keywords: Acute myocardial infarction; Non-ST Segment Elevation MI; ST-Elevation Myocardial Infarction; Dual antiplatelet therapy; Helicobacter pylori; Screening; Upper gastrointestinal bleeding; Urea breath test
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Helicobacter Screening (Experimental): All patients with confirmed MI (both STEMI and NSTEMI) will be tested for Hp infection with bedside UBT.
  Interventions: Diagnostic Test: Helicobacter Pylori screening by UBT

INTERVENTIONS:
Diagnostic Test: Helicobacter Pylori screening by UBT — The UBT is based on the fact that Hp produces urease, which catalyzes the urea molecule into ammonia (NH3) and carbon dioxide (CO2). After fasting for six hours prior to testing, the patient swallows a C13 Urea tablet or solution and waits. After 10 minutes, the patient exhales and breath is collected (tube, bag or breath card). The production of 13CO2 is measured by a desktop analyzer (infrared mass spectrometry) and Hp diagnosis is made based on previously established cut-off levels for Hp infection.

SUMMARY:
The aim of this study is to determine the prevalence of Helicobacter pylori (Hp) infection in patients with myocardial infarction (MI). This is performed to establish the feasibility of a large trial examining whether systematic screening for and subsequent eradication therapy significantly reduces the risk of hospitalization for upper gastrointestinal (GI) bleeding in patients after MI.

DETAILED DESCRIPTION:
Despite progressively reduced mortality over the last decades, cardiovascular disease remains the most common cause of death in both men and women in Sweden and the world. In addition to early revascularization therapy, potent antithrombotic therapy is the basis for the reduction in cardiovascular events, however, at a price of increased risk of bleeding, typically upper gastrointestinal bleeding (UGIB) that result in substantial morbidity, mortality, and medical care cost. Risk factors for UGIB include high age, male sex, renal failure, and a chronic bacterial infection caused by Helicobacter pylori (Hp), the latter being the only treatable. H. pylori infection causes both acute and chronic gastritis with ulcerative and erosive lesions, peptic ulcer disease (both duodenal and gastric ulcers) and, less commonly, gastric cancer and mucosa-associated lymphoid tissue (MALT) lymphoma. Concomitant anticoagulation or antithrombotic therapy aggravates the risk for bleeding, 2-fold with low dose aspirin, up to 7-fold with dual antiplatelet therapy, which today is standard treatment for 12 months post MI.

Non-invasive screening for Hp can be performed easily with high accuracy by urea breath or stool test. If found positive, eradication by triple therapy is well established and recommended in risk individuals and believed to reverse the bleeding risk almost completely.

Hp screening in a current MI population has to our knowledge never been performed. Thus, it remains unknown if systematic screening and subsequent eradication therapy significantly reduces the risk of bleeding and improves prognosis.

The HELicobacter Pylori Screening in Patients With Acute Myocardial Infarction (HELP) pilot study is a multicenter, single group, open-label, clinical trial evaluating the prevalence of Hp in patients hospitalized with acute MI.

All patients at participating sites during the inclusion period, with MI diagnosis defined as International Classification of Diseases (ICD) codes I21 or I22, and age≥18 years, are eligible for enrollment. After written informed consent eligible patients will be tested for Hp infection with a bedside urea breath test (UBT) incorporated into MI routine care during the hospitalization period.

The UBT is based on the fact that Hp produces urease, which catalyzes the urea molecule into ammonia (NH3) and carbon dioxide (CO2). After fasting for six hours prior to testing, the patient swallows a C13 Urea tablet or solution and waits. After 10 minutes, the patient exhales and breath is collected (tube, bag or breath card). The production of 13CO2 is measured by a desktop analyzer (infrared mass spectrometry) and Hp diagnosis is made based on previously established cut-off levels for Hp infection.

In patients tested positive, standard triple eradication therapy according to the national society of gastroenterology guidelines will be prescribed at the caring physician's discretion.

Control of successful Hp eradication therapy according to guidelines with either UBT or Hp-antigen in feces 6 weeks after completed eradication therapy is recommended to the treating physician.

Baseline characteristics and data about the in-hospital period (medication, procedures, complications, laboratory results) will be collected from the Swedish Web System for Enhancement and Development of Evidence-based Care in Heart Disease Evaluated According to Recommended Therapies (SWEDEHEART) registry. For patients with acute MI, 106 variables are registered, including demographics, risk factors, past medical history, medical treatment before admission, electrocardiographic changes, echocardiography, biochemical markers, other clinical features and investigations, medical treatment in hospital, interventions, hospital outcome, discharge diagnoses and discharge-medications.

Primary objective of this pilot study is to determine the prevalence of Hp infection in patients with MI.

The secondary objective is to determine the feasibility of a large clinical trial on whether systematic screening for Hp and subsequent eradication therapy in patients after MI reduces UGIB and cardiovascular events.

The tertiary objective is to map if the cardiovascular risk profile differs in patients that are Hp negative and Hp positive, respectively.

All-cause death within 30 days will be obtained from the Swedish population registry, including the vital status of all Swedish residence. SWEDEHEART is linked to the Swedish population registry every month.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 myocardial infarction (both STEMI and NSTEMI)

Exclusion Criteria:

* Only concerning UBT (Patients after gastric surgery, with acute gastrointestinal bleeding, suspected gastric infection, or known atrophic gastritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hp | Baseline
  Prevalence of Hp assessed by UBT

SECONDARY OUTCOMES:
Baseline characteristics according to Hp screening result | Baseline
  Comparison of baseline characteristics according to Hp screening result (positive/negative)
Baseline characteristics according to Hp screening result and infarct type | Baseline
  Comparison of baseline characteristics according to Hp screening result (positive/negative) stratified by infarct type
Baseline characteristics according to Hp screening result, infarct type and concomitant therapy | Baseline
  Comparison of baseline characteristics according to Hp screening result (positive/negative) stratified by infarct type and concomitant therapy (PPI, antibiotics)
All-cause mortality | 30 days
  All-cause mortality in Hp screened Mi patients according to screening status

CONTACTS AND LOCATIONS:
Overall Officials: Robin Hofmann, MD, PhD, Principal Investigator — Karolinska Institutet, Södersjukhuset
Locations (2):
- Sweden (2):
  - Karolinska University Hospital Huddinge, Huddinge
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laine L. CLINICAL PRACTICE. Upper Gastrointestinal Bleeding Due to a Peptic Ulcer. N Engl J Med. 2016 Jun 16;374(24):2367-76. doi: 10.1056/NEJMcp1514257. No abstract available. PMID 27305194
- [Result] Sarri GL, Grigg SE, Yeomans ND. Helicobacter pylori and low-dose aspirin ulcer risk: A meta-analysis. J Gastroenterol Hepatol. 2019 Mar;34(3):517-525. doi: 10.1111/jgh.14539. Epub 2018 Dec 17. PMID 30408229
- [Result] Chan FK, Ching JY, Suen BY, Tse YK, Wu JC, Sung JJ. Effects of Helicobacter pylori infection on long-term risk of peptic ulcer bleeding in low-dose aspirin users. Gastroenterology. 2013 Mar;144(3):528-35. doi: 10.1053/j.gastro.2012.12.038. Epub 2013 Jan 16. PMID 23333655
- [Result] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Result] Dzierzanowska-Fangrat K, Lehours P, Megraud F, Dzierzanowska D. Diagnosis of Helicobacter pylori infection. Helicobacter. 2006 Oct;11 Suppl 1:6-13. doi: 10.1111/j.1478-405X.2006.00423.x. PMID 16925605